CLINICAL TRIAL: NCT00197275
Title: Demonstrate Lot-to-lot Consistency of Final Production Method of GSK Biologicals' Hib-MenAC Vaccine Mixed Extemporaneously With Tritanrix™-HepB & Demonstrate Its Non-inferiority vs Tritanrix™-HepB/Hiberix™ in Healthy Infants at 2, 4 and 6 Months
Brief Title: Lot-to-lot Consistency of Tritanrix™-HepB/Hib-MenAC & Its Non-inferiority vs Tritanrix™-HepB/Hiberix™ in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 104733
Record Dates: First submitted 2005-09-19; First posted 2005-09-20 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Tetanus; Hepatitis B; Haemophilus Influenzae Type b; Whole Cell Pertussis; Diphtheria
Keywords: Haemophilus influenzae type b; diphtheria; tetanus; Prophylaxis diphtheria; pertussis; hepatitis B; meningococcal serogroups A & C diseases
MeSH Terms: conditions — Tetanus; Hepatitis B; Haemophilus Infections; Diphtheria; Whooping Cough

INTERVENTIONS:
Biological: Hib-MenAC mixed with Tritanrix™-HepB

SUMMARY:
The primary purpose of this study is to demonstrate the lot-to-lot consistency of 3 production lots of GSK Biologicals' Hib-MenAC (Haemophilus influenzae type b and meningococcal serogroups A and C) vaccine when reconstituted with Tritanrix™-HepB (diphtheria, tetanus, pertussis, and hepatitis B) vaccine and administered as a single injection.

DETAILED DESCRIPTION:
The study is double blind. However the active control vaccine Tritanrix™-HepB/Hiberix™ will be administered in a single-blind manner. Blood samples will be collected for immunogenicity analyses. GSK Biologicals' OPV vaccine will be administered concomitantly with the study vaccines at 2, 4 and 6 months of age according to local country regulation. The study will last approximately 5 months per subject

ELIGIBILITY:
Inclusion criteria:

* healthy male or female, between, and including, 56 and 83 days of age.
* Born after a gestation period between 36 and 42 weeks
* Birth dose of hepatitis B vaccine within the first 72 hours of life

Exclusion criteria:

* planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of study vaccine, or planned administration during the study period.
* Bacille Calmette-Guérin (BCG) vaccine received after the first 2 weeks of life.
* History of OR previous vaccination against OR known exposure since birth to diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b and/or meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* A family history of congenital or hereditary immunodeficiency
* History of any neurologic disorders or seizures
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine

Ages: 56 Days to 83 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800
Dates: Start 2006-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Immune response 1 month post dose 3 (SBA-MenA/C titers ≥ 1:8, anti-PRP ≥ 0.15 µg/ml, -diphtheria ≥ 0.1 IU/ml (ELISA) OR ≥ 0.016 IU/ml (Vero-cell test), -tetanus ≥ 0.1 IU/ml, -HB concentration ≥ 10 mIU/ml, vaccine response to Bordetella pertus

SECONDARY OUTCOMES:
Antibody conc or titer, seroprot, seropos and/or vacc response to all antigens administered (Prior to dose 1, 2 m after dose 2 & 1m after dose 3). After each dose: Solicited (d 0-3, local/general), unsolicited (d 0-30) symptoms. During whole study: SAEs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Guignard A, Haguinet F, Wery S, Kerdpanich P. Prevalence and Persistence of Maternal Dengue Neutralizing Antibodies in Infants From Central and Southern Thailand: A Retrospective Cohort Study. Asia Pac J Public Health. 2019 May;31(4):288-295. doi: 10.1177/1010539519853396. PMID 31307216
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104733 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104733 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104733 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104733 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104733 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104733 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register